CLINICAL TRIAL: NCT02087046
Title: A Clinical Evaluation of the Advanced Neuromodulation System (ANS) Totally Implantable Deep Brain Stimulation System for the Suppression of Tremor in the Upper Extremities of Patients With Essential Tremor.
Brief Title: Deep Brain Stimulation (DBS) for the Suppression of Tremor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-04-02
Record Dates: First submitted 2014-03-12; First posted 2014-03-14 (Estimated); Results first posted 2021-02-26 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Tremor; Action Tremor; Essential Tremor; Tremor, Limb
MeSH Terms: conditions — Tremor; Essential Tremor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stimulation (Other): ANS Totally Implantable Deep Brain Stimulation System
  Interventions: Device: ANS Totally Implantable Deep Brain Stimulation System

INTERVENTIONS:
Device: ANS Totally Implantable Deep Brain Stimulation System — ANS Totally Implantable Deep Brain Stimulation System will be implanted in the VIM nucleus of the thalamus

SUMMARY:
The purpose of the proposed study is to demonstrate the safety and efficacy of the ANS Totally Implantable Deep Brain Stimulation System in the VIM nucleus of the thalamus implanted for the treatment of tremor due to essential tremor.

This study will be included in the Pre-Market Approval Application to support the safety of this device in use.

DETAILED DESCRIPTION:
This study is designed as a prospective, multi-centered study for 365 days in duration from device implantation. A maximum of 12 sites will enroll 160 patients.

Each patient will be screened and then undergo a baseline evaluation followed by unilateral or bilateral implantation of the DBS system. During the implantation procedure, each patient will undergo a trial of stimulation in the operating room. The device may be internalized after a successful intra-operative trial or at a later surgery (no later than 4 weeks after initial lead placement). If the device is not activated immediately postsurgery, the patient may return to the clinic to determine optimum stimulation programming. Device programming will be optimized in as many visits as necessary following implantation. The day that the device is fully implanted will be classified as "Day 0" for each patient.

After "Day 0" the patient will return to clinic for evaluations at, Day 90 (±14 days), and Day 180 (±14 days) and Day 365 (approximately 12 months ± 30 days after Day 0). These evaluations consist of the CRST, the QUEST, the SF36, Patient and caregiver Global Ratings and the Patient Satisfaction Rating.

At Baseline and Day 180, the CRST evaluation session will be video recorded for analysis by an independent evaluator unaware of the functioning of the device. Additionally, at the Day 180 visit, the physician will have the option to provide the patient with amplitude control. A comparison of measures within the same person from pre-treatment to post-treatment will be performed. Also, pre-treatment and post-treatment group means and standard deviations will be determined.

Patients completed follow-up visits as part of the original protocol (C-04-02) for one year (or in some cases longer if patient was bilaterally implanted) and continued to complete additional visits as part of the Long-Term Follow-up protocol (C-06-03) for up to 5 years post implant.

ELIGIBILITY:
Inclusion criteria:

1. Patient or authorized representative has signed an informed consent.
2. Patient is over 18 years of age.
3. Patient is diagnosed with essential tremor for at least 3 years.
4. Patient has a disabling medical-refractory upper extremity tremor with no evidence of supraspinal central nervous system disease or injury (tremor not adequately controlled by medications for at least three (3) months before implant).
5. Patient has a postural or kinetic tremor severity score of at least 3 out of 4 in the extremity intended for treatment on the Fahn-Tolosa-Marin Clinical Rating Scale for Tremor.
6. Patient will maintain a constant dose of anti-tremor medication indicated as best medical management for one (1) month prior to enrollment in study.
7. Patient is available for appropriate follow-up times for the length of the study.

Exclusion criteria:

1. Patient is not surgical candidate;
2. Patient has other clinically or medically significant disease;
3. Patient has any neurological injury or disease other than essential tremor;
4. Patient has any condition requiring repeated MRI scans;
5. Patient has any condition requiring diathermy;
6. Patients on anticoagulant medications;
7. Patient has untreated clinically significant depression;
8. Patient has had an electrical or electromagnetic implant (cochlear prosthesis, pacemaker etc);
9. Patient has had a prior thalamotomy or surgical ablation procedure in either side of the brain;
10. Patient has dementia interfering with their ability to co-operate or comply with study requirements or comprehend the informed consent (mini-mental exam score <24);
11. Patient abuses drugs or alcohol;
12. Patient has had botulinum toxin injections in the six (6) months prior to enrollment;
13. Patient has a history of cranial surgery;
14. Patient has a history of seizures;
15. Patient has any metallic implants that may interfere with the functioning of the device (e.g. aneurysm clips);
16. Patient has a history of stimulation intolerance in any area of the body;
17. Patient is a female of child bearing potential with a positive urine pregnancy test or not using adequate contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2005-10; Primary Completion 2014-04 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Karst, Study Director — Abbott
Locations (12):
- United States (12):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Loma Linda University School of Medicine, Loma Linda, California
  - Pacific Hills Neurosurgery Medical Group, Pasadena, California
  - University of San Francisco, San Francisco, California
  - University of Florida, Gainesville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Oakwood Hospital, Dearborn, Michigan
  - Columbia University Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Vanderbilt University, Nashville, Tennessee
  - Neurology Specialists of Dallas, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 127 patients were enrolled from 12 investigational sites and implanted with the study device. The first patient was implanted with the SJM DBS Systems on 21 October, 2005. Of the 127 implanted subjects, 80 received unilateral implants and the remaining 47 patients received bilateral implants.
Pre-assignment Details: Of the 150 subjects who were screened, 23 subjects were excluded from implantation due to inclusion or exclusion criteria, or the patient's decision to discontinue before surgery.
Groups:
- Stimulation: ANS Totally Implantable Deep BrainStimulation System: ANS Totally Implantable Deep BrainStimulation System will be implanted in the VIM nucleus of the thalamus
Period: Overall Study
Arm/Group | Stimulation
Started | 127
Primary Endpoint | 121
Completed | 116
Not Completed | 11
Not completed — Adverse Event | 4
Not completed — Death | 1
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Stimulation
Number analyzed (Participants) | 127
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58
  Male | 69
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 124
  African American | 1
  Hispanic | 2
Region of Enrollment [Number; unit: participants]
  United States | 127
Years since onset of tremor [Mean (Standard Deviation); unit: years] | 29.1 (17.4)
Years since initial diagnosis of ET [Mean (Standard Deviation); unit: years] | 14.8 (11.8)

OUTCOME MEASURES:

1. Primary Outcome: Primary Efficacy Endpoint: Difference in the Postural Tremor Score of the Target Limb Between Stimulation On and Stimulation Off, As Assessed by the Blind Reviewer
Description: The Fahn, Tolosa, Marin Tremor Rating Scale (referred to as the CRST), is a rating tool to assess the severity of postural, isometric, kinetic and task specific tremor in the dominant and non-dominant sides of the head, trunk and limbs of patients with ET. The CRST utilizes a 0 to 4 point scale where 0 indicates non-symptomatic (normal) and 4 indicates the most severe rating of the patient's tremor symptoms.
Time Frame: Day 180
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stimulation
Number analyzed (Participants) | 76
units on a scale
  Stimulation Off | 2.09 (1.07)
  Stimulation On | 0.84 (0.83)
  Mean Difference | -1.25 (1.26)

2. Primary Outcome: Primary Safety Endpoint: Percentage of Participants With Device-related or Procedure Related Adverse Events
Description: Percentage of device-related or procedure related adverse events will be assessed within 6 months following the initial unilateral implant. All such adverse events will be counted for 180 days following surgery or until the day of the second implant, which ever comes first.
Time Frame: Within 180 days following the initial implant
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Number; unit: percentage of participants
Arm/Group | Stimulation
Number analyzed (Participants) | 127
percentage of participants | 31.5

3. Secondary Outcome: Clinical Rating Scale for Tremor (CRST) Evaluation- Mean Target Limb Severity Score, As Assessed by the Site Physician
Description: as for outcome 1
Time Frame: Baseline
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stimulation
Number analyzed (Participants) | 122
score on a scale | 3.10 (0.62)

4. Secondary Outcome: Clinical Rating Scale for Tremor (CRST) Evaluation- Mean Target Limb Severity Score, As Assessed by the Site Physician
Description: as for outcome 1
Time Frame: Day 90
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stimulation
Number analyzed (Participants) | 121
score on a scale
  Stimulation Off | 2.41 (0.98)
  Stimulation On | 0.75 (0.78)
  Mean Difference | -1.66 (1.07)

5. Secondary Outcome: Clinical Rating Scale for Tremor (CRST) Evaluation- Mean Target Limb Severity Score, As Assessed by the Site Physician
Description: as for outcome 1
Time Frame: Day 180
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stimulation
Number analyzed (Participants) | 118
score on a scale
  Stimulation Off | 2.41 (0.96)
  Stimulation On | 0.67 (0.70)
  Mean Difference | -1.74 (1.10)

6. Secondary Outcome: Clinical Rating Scale for Tremor (CRST) Evaluation- Mean Target Limb Severity Score, As Assessed by the Site Physician
Description: as for outcome 1
Time Frame: Day 365
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stimulation
Number analyzed (Participants) | 112
score on a scale
  Stimulation Off | 2.55 (1.12)
  Stimulation On | 0.62 (0.79)
  Mean Difference | -1.94 (1.16)

7. Secondary Outcome: Clinical Rating Scale for Tremor (CRST) Evaluation- Target Limb Responder Analysis, As Assessed by the Site Physician
Description: The Fahn, Tolosa, Marin Tremor Rating Scale (referred to as the CRST), is a rating tool to assess the severity of postural, isometric, kinetic and task specific tremor in the dominant and non-dominant sides of the head, trunk and limbs of patients with ET. The CRST utilizes a 0 to 4 point scale where 0 indicates non-symptomatic (normal) and 4 indicates the most severe rating of the patient's tremor symptoms.
  During responder analysis, a 2-point reduction in kinetic tremor or postural tremor between stimulation Off and stimulation On show an improvement in activities of daily living was considered a response, was also performed using the site physician's ratings.
Time Frame: Day 90
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Stimulation
Number analyzed (Participants) | 121
Participants
  Between Stimulation OFF and Stimulation ON | 67
  Between Baseline and Stimulation ON | 98

8. Secondary Outcome: Clinical Rating Scale for Tremor (CRST) Evaluation- Target Limb Responder Analysis, As Assessed by the Site Physician
Description: as for outcome 7
Time Frame: Day 180
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Stimulation
Number analyzed (Participants) | 118
Participants
  Between Stimulation OFF and Stimulation ON | 69
  Between Baseline and Stimulation ON | 98

9. Secondary Outcome: Clinical Rating Scale for Tremor (CRST) Evaluation- Target Limb Responder Analysis, As Assessed by the Site Physician
Description: as for outcome 7
Time Frame: Day 365
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Stimulation
Number analyzed (Participants) | 112
Participants
  Between Stimulation OFF and Stimulation ON | 72
  Between Baseline and Stimulation ON | 97

10. Secondary Outcome: Clinical Rating Scale for Tremor (CRST) Evaluation- Mean Handwriting for Target Side Severity Score, As Assessed by the Site Physician
Description: The Fahn, Tolosa, Marin Tremor Rating Scale (referred to as the CRST), is a rating tool to assess the severity of postural, isometric, kinetic and task specific tremor in the dominant and non-dominant sides of the head, trunk and limbs of patients with ET. The CRST utilizes a 0 to 4 point scale where 0 indicates non-symptomatic (normal) and 4 indicates the most severe rating of the patient's tremor symptoms.
  The site physician will evaluate the patient's handwriting according to the CRST (scale 0-4).
Time Frame: Baseline
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stimulation
Number analyzed (Participants) | 122
score on a scale | 2.66 (0.97)

11. Secondary Outcome: Clinical Rating Scale for Tremor (CRST) Evaluation- Mean Handwriting for Target Side Severity Score, As Assessed by the Site Physician
Description: as for outcome 10
Time Frame: Day 90
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stimulation
Number analyzed (Participants) | 121
score on a scale
  Stimulation Off | 2.18 (1.14)
  Stimulation On | 0.93 (0.91)
  Mean Difference | -1.25 (0.95)

12. Secondary Outcome: Clinical Rating Scale for Tremor (CRST) Evaluation- Mean Handwriting for Target Side Severity Score, As Assessed by the Site Physician
Description: as for outcome 10
Time Frame: Day 180
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Stimulation: ANS Totally Implantable Deep BrainStimulation System: ANS Totally Implantable Deep BrainStimulation System will be implanted in theVIM nucleus of the thalamus
Arm/Group | Stimulation
Number analyzed (Participants) | 117
score on a scale
  Stimulation Off | 2.22 (1.08)
  Stimulation On | 0.91 (0.89)
  Mean Difference | -1.32 (1.06)

13. Secondary Outcome: Clinical Rating Scale for Tremor (CRST) Evaluation- Mean Handwriting for Target Side Severity Score, As Assessed by the Site Physician
Description: as for outcome 10
Time Frame: Day 365
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stimulation
Number analyzed (Participants) | 110
score on a scale
  Stimulation Off | 2.32 (1.14)
  Stimulation On | 0.90 (0.87)
  Mean Difference | -1.42 (1.10)

14. Secondary Outcome: Clinical Rating Scale for Tremor (CRST) Evaluation- Mean Handwriting for Target Side Severity Score, As Assessed by the Blind Reviewer
Description: The Fahn, Tolosa, Marin Tremor Rating Scale (referred to as the CRST), is a rating tool to assess the severity of postural, isometric, kinetic and task specific tremor in the dominant and non-dominant sides of the head, trunk and limbs of patients with ET. The CRST utilizes a 0 to 4 point scale where 0 indicates non-symptomatic (normal) and 4 indicates the most severe rating of the patient's tremor symptoms.
  The blind reviewer will evaluate the patient's handwriting according to the CRST (scale 0-4).
Time Frame: Day 180
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stimulation
Number analyzed (Participants) | 58
score on a scale
  Stimulation Off | 1.69 (1.10)
  Stimulation On | 0.62 (0.72)
  Mean Difference | -1.07 (1.06)

15. Secondary Outcome: Clinical Rating Scale for Tremor (CRST) Evaluation- Mean Pouring From Target Side Severity Scores, As Assessed by the Site Physician
Description: The Fahn, Tolosa, Marin Tremor Rating Scale (referred to as the CRST), is a rating tool to assess the severity of postural, isometric, kinetic and task specific tremor in the dominant and non-dominant sides of the head, trunk and limbs of patients with ET. The CRST utilizes a 0 to 4 point scale where 0 indicates non-symptomatic (normal) and 4 indicates the most severe rating of the patient's tremor symptoms.
  The site physician will evaluate the patient's pouring ability according to the CRST
Time Frame: Baseline
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stimulation
Number analyzed (Participants) | 122
score on a scale | 2.56 (0.98)

16. Secondary Outcome: Clinical Rating Scale for Tremor (CRST) Evaluation-Mean Pouring From Target Side Severity Scores, As Assessed by the Site Physician
Description: as for outcome 15
Time Frame: Day 90
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stimulation
Number analyzed (Participants) | 121
score on a scale
  Stimulation Off | 2.25 (1.14)
  Stimulation On | 0.68 (0.90)
  Mean Difference | -1.57 (1.17)

17. Secondary Outcome: Clinical Rating Scale for Tremor (CRST) Evaluation- Mean Pouring From Target Side Severity Scores, As Assessed by the Site Physician
Description: as for outcome 15
Time Frame: Day 180
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stimulation
Number analyzed (Participants) | 118
score on a scale
  Stimulation Off | 2.08 (1.19)
  Stimulation On | 0.57 (0.76)
  Mean Difference | -1.52 (1.11)

18. Secondary Outcome: Clinical Rating Scale for Tremor (CRST) Evaluation-Mean Pouring From Target Side Severity Scores, As Assessed by the Site Physician
Description: as for outcome 15
Time Frame: Day 365
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stimulation
Number analyzed (Participants) | 112
score on a scale
  Stimulation Off | 2.16 (1.31)
  Stimulation On | 0.62 (0.91)
  Mean Difference | -1.54 (1.06)

19. Secondary Outcome: Clinical Rating Scale for Tremor (CRST) Evaluation- Pouring Ability From Target Side Severity Scores, As Assessed by the Blind Reviewer
Description: The Fahn, Tolosa, Marin Tremor Rating Scale (referred to as the CRST), is a rating tool to assess the severity of postural, isometric, kinetic and task specific tremor in the dominant and non-dominant sides of the head, trunk and limbs of patients with ET. The CRST utilizes a 0 to 4 point scale where 0 indicates non-symptomatic (normal) and 4 indicates the most severe rating of the patient's tremor symptoms.
  The blind reviewer will evaluate the patient's pouring ability according to the CRST
Time Frame: Day 180
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stimulation
Number analyzed (Participants) | 50
score on a scale
  Stimulation Off | 1.56 (1.13)
  Stimulation On | 0.70 (0.86)
  Mean Difference | -0.86 (1.09)

20. Secondary Outcome: Clinical Rating Scale for Tremor (CRST) Evaluation- Mean Total Motor Score, As Assessed by the Site Physician
Description: The Fahn, Tolosa, Marin Tremor Rating Scale (referred to as the CRST), is a rating tool to assess the severity of postural, isometric, kinetic and task specific tremor in the dominant and non-dominant sides of the head, trunk and limbs of patients with ET. The CRST utilizes a 0 to 4 point scale where 0 indicates non-symptomatic (normal) and 4 indicates the most severe rating of the patient's tremor symptoms.
  The motor score adds together all responses to the tremor assessment for questions 1-9 of the CRST (whether or not the specific side is being treated).
Time Frame: Baseline
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stimulation
Number analyzed (Participants) | 122
score on a scale | 16.9 (5.9)

21. Secondary Outcome: Clinical Rating Scale for Tremor (CRST) Evaluation- Mean Total Motor Score, As Assessed by the Site Physician
Description: as for outcome 20
Time Frame: Day 90
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stimulation
Number analyzed (Participants) | 119
score on a scale
  Stimulation Off | 13.1 (6.8)
  Stimulation On | 7.9 (4.8)
  Mean Difference | -5.2 (3.8)

22. Secondary Outcome: Clinical Rating Scale for Tremor (CRST) Evaluation- Mean Total Motor Score, As Assessed by the Site Physician
Description: as for outcome 20
Time Frame: Day 180
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stimulation
Number analyzed (Participants) | 116
score on a scale
  Stimulation Off | 13.6 (6.9)
  Stimulation On | 7.4 (4.1)
  Mean Difference | -6.2 (4.8)

23. Secondary Outcome: Clinical Rating Scale for Tremor (CRST) Evaluation- Mean Total Motor Score, As Assessed by the Site Physician
Description: as for outcome 20
Time Frame: Day 365
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stimulation
Number analyzed (Participants) | 112
score on a scale
  Stimulation Off | 14.6 (8.8)
  Stimulation On | 7.2 (5.0)
  Mean Difference | -7.4 (6.6)

24. Secondary Outcome: Clinical Rating Scale for Tremor (CRST) Evaluation- Activity of Daily Living Score, As Assessed by the Site Physician
Description: The Fahn, Tolosa, Marin Tremor Rating Scale (referred to as the CRST), is a rating tool to assess the severity of postural, isometric, kinetic and task specific tremor in the dominant and non-dominant sides of the head, trunk and limbs of patients with ET. The CRST utilizes a 0 to 4 point scale where 0 indicates non-symptomatic (normal) and 4 indicates the most severe rating of the patient's tremor symptoms.
  The activity of daily living score adds together all responses to questions 15-21 of the CRST.
Time Frame: Baseline
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stimulation
Number analyzed (Participants) | 123
score on a scale | 16.3 (3.9)

25. Secondary Outcome: Clinical Rating Scale for Tremor (CRST) Evaluation- Activity of Daily Living Score, As Assessed by the Site Physician
Description: as for outcome 24
Time Frame: Day 90
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stimulation
Number analyzed (Participants) | 122
score on a scale
  Stimulation Off | 13.8 (6.1)
  Stimulation On | 5.0 (4.7)
  Mean Difference | -8.8 (5.5)

26. Secondary Outcome: Clinical Rating Scale for Tremor (CRST) Evaluation- Activity of Daily Living Score, As Assessed by the Site Physician
Description: as for outcome 24
Time Frame: Day 180
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stimulation
Number analyzed (Participants) | 118
score on a scale
  Stimulation Off | 14.3 (6.2)
  Stimulation On | 5.2 (4.6)
  Mean Difference | -9.1 (6.1)

27. Secondary Outcome: Clinical Rating Scale for Tremor (CRST) Evaluation- Activity of Daily Living Score, As Assessed by the Site Physician
Description: as for outcome 24
Time Frame: Day 365
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stimulation
Number analyzed (Participants) | 107
score on a scale
  Stimulation Off | 14.7 (6.5)
  Stimulation On | 4.6 (4.7)
  Mean Difference | -10.0 (5.4)

28. Secondary Outcome: Clinical Rating Scale for Tremor (CRST) Evaluation-Bilateral Stimulation, As Assessed by the Site Physician
Description: The Fahn, Tolosa, Marin Tremor Rating Scale (referred to as the CRST), is a rating tool to assess the severity of postural, isometric, kinetic and task specific tremor in the dominant and non-dominant sides of the head, trunk and limbs of patients with ET. The CRST utilizes a 0 to 4 point scale where 0 indicates non-symptomatic (normal) and 4 indicates the most severe rating of the patient's tremor symptoms.
  For those patients that had bilateral stimulation, the site physician will evaluate the patient's non-target side after 180 days of bilateral stimulation.
Time Frame: Baseline
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stimulation
Number analyzed (Participants) | 39
score on a scale | 2.82 (0.76)

29. Secondary Outcome: Clinical Rating Scale for Tremor (CRST) Evaluation-Bilateral Stimulation, As Assessed by the Site Physician
Description: as for outcome 28
Time Frame: Following 180 days of stimulation
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stimulation
Number analyzed (Participants) | 39
score on a scale
  Stimulation Off | 2.67 (0.87)
  Stimulation On | 0.95 (0.89)
  Mean Difference | -1.72 (1.00)

30. Secondary Outcome: Clinical Rating Scale for Tremor (CRST) Evaluation-Non-Target Limb Severity Scores, As Assessed by the Site Physician
Description: The Fahn, Tolosa, Marin Tremor Rating Scale (referred to as the CRST), is a rating tool to assess the severity of postural, isometric, kinetic and task specific tremor in the dominant and non-dominant sides of the head, trunk and limbs of patients with ET. The CRST utilizes a 0 to 4 point scale where 0 indicates non-symptomatic (normal) and 4 indicates the most severe rating of the patient's tremor symptoms.
  For those patients that had bilateral stimulation, the site physician will evaluate the patient's non-target side after 180 days with only the second side system On
Time Frame: Baseline
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stimulation
Number analyzed (Participants) | 37
score on a scale | 2.84 (0.80)

31. Secondary Outcome: Clinical Rating Scale for Tremor (CRST) Evaluation-Non-Target Limb Severity Scores, As Assessed by the Site Physician
Description: as for outcome 30
Time Frame: Following 180 days of stimulation
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stimulation
Number analyzed (Participants) | 37
score on a scale
  Stimulation Off | 2.73 (0.90)
  Stimulation On | 1.11 (1.07)
  Mean Difference | -1.62 (1.06)

32. Secondary Outcome: Quality of Life in Essential Tremor (QUEST): Overall Summary Index
Description: The QUEST questionnaire consists of 30 items, which are rated from 0 to 4, corresponding to the frequency (from never to always). Those 30 items assess how tremor impacts a function or how it can be associated with feelings or attitudes. The 30 items contribute to five sub scales (number of items contributing to each scale in parentheses): Physical/ADL (9), Psychosocial (9), Communication (3), Hobbies/Leisure (3), and Work/Finances (6). The score on each sub scale is expressed as a percentage of the total score possible, with a higher score indicating greater dissatisfaction with that domain of QOL. As the scores were expressed as percentages, if a question was unanswered it was excluded and percentages were calculated based on the remaining answers. A total or quest summary index (QSI) was computed by calculating the mean of the five scales. Maximal score of 100 indicates worse quality of life, while minimal score 0 corresponds to best quality of life.
Time Frame: Baseline
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stimulation
Number analyzed (Participants) | 123
score on a scale | 49.1 (12.6)

33. Secondary Outcome: Change From Baseline for Quality of Life in Essential Tremor (QUEST): Overall Summary Index
Description: as for outcome 32
Time Frame: Day 90
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stimulation
Number analyzed (Participants) | 122
score on a scale
  Summary Index Mean | 33.1 (16.8)
  Mean Change in Summary Index | -16.0 (15.5)

34. Secondary Outcome: Change From Baseline for Quality of Life in Essential Tremor (QUEST): Overall Summary Index
Description: as for outcome 32
Time Frame: Day 180
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stimulation
Number analyzed (Participants) | 118
score on a scale
  Summary Index Mean | 33.0 (16.2)
  Mean Change in Summary Index | -15.9 (16.9)

35. Secondary Outcome: Change From Baseline for Quality of Life in Essential Tremor (QUEST): Overall Summary Index
Description: as for outcome 32
Time Frame: Day 365
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stimulation
Number analyzed (Participants) | 110
score on a scale
  Summary Index | 30.9 (16.4)
  Mean Change in Summary Index | -18.0 (15.4)

36. Secondary Outcome: SF36 Components and Individual Domains
Description: The SF-36 questionnaire is a measure of health status with 36 items across 8 domains. The eight domains are separated into two summary scores of four domains, the physical component summary (PCS) and mental component summary (MCS). The SF-36 score is transformed into a scale of 0-100, with 100 indicating no disability. PCS and MCS are scaled in comparison to population norms to reflect a mean of 50 and standard deviation of 10 for the general population of the United States.
Time Frame: Baseline
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stimulation
Number analyzed (Participants) | 123
score on a scale
  Physical Component Summary | 45.62 (9.49)
  Mental Component Summary | 50.11 (10.9)

37. Secondary Outcome: SF36 Components and Individual Domains
Description: as for outcome 36
Time Frame: Day 90
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stimulation
Number analyzed (Participants) | 122
score on a scale
  Physical Component Summary | 47.21 (8.45)
  Mental Component Summary | 52.71 (8.07)

38. Secondary Outcome: SF36 Components and Individual Domains
Description: as for outcome 36
Time Frame: Day 180
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stimulation
Number analyzed (Participants) | 117
score on a scale
  Physical Component Summary | 46.82 (9.94)
  Mental Component Summary | 51.85 (9.51)

39. Secondary Outcome: SF36 Components and Individual Domains
Description: as for outcome 36
Time Frame: Day 365
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stimulation
Number analyzed (Participants) | 108
score on a scale
  Physical Component Summary | 45.6 (9.79)
  Mental Component Summary | 52.21 (10.15)

40. Secondary Outcome: Global Assessment Scores by Examiner
Description: Global outcome measures are a self-rated questionnaire that measures a global assessment of the patient quality of life and the examiner's interpretation of the patient's quality of life.
Time Frame: Baseline
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Stimulation
Number analyzed (Participants) | 122
Participants
  No disability | 0
  Mild disability | 2
  Moderate disability | 35
  Marked disability | 68
  Severe disability | 17

41. Secondary Outcome: Global Assessment Scores by Examiner
Description: as for outcome 40
Time Frame: Day 90
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Stimulation
Number analyzed (Participants) | 122
Participants
  No disability | 28
  Mild disability | 66
  Moderate disability | 21
  Marked disability | 5
  Severe disability | 2

42. Secondary Outcome: Global Assessment Scores by Examiner
Description: as for outcome 40
Time Frame: Day 180
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Stimulation
Number analyzed (Participants) | 118
Participants
  No disability | 31
  Mild disability | 57
  Moderate disability | 25
  Marked disability | 5
  Severe disability | 0

43. Secondary Outcome: Global Assessment Scores by Examiner
Description: as for outcome 40
Time Frame: Day 365
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Stimulation
Number analyzed (Participants) | 110
Participants
  No disability | 36
  Mild disability | 55
  Moderate disability | 14
  Marked disability | 4
  Severe disability | 1

44. Secondary Outcome: Global Assessment by Caregiver
Description: Global outcome measures are a self-rated questionnaire that measures a global assessment of the patient quality of life and the caregiver's interpretation of the patient's quality of life
Time Frame: Baseline
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Stimulation
Number analyzed (Participants) | 68
Participants
  No disability | 0
  Mild disability | 2
  Moderate disability | 15
  Marked disability | 32
  Severe disability | 19

45. Secondary Outcome: Global Assessment by Caregiver
Description: as for outcome 44
Time Frame: Day 90
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Stimulation
Number analyzed (Participants) | 72
Participants
  No disability | 19
  Mild disability | 33
  Moderate disability | 13
  Marked disability | 5
  Severe disability | 2

46. Secondary Outcome: Global Assessment by Caregiver
Description: as for outcome 44
Time Frame: Day 180
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Stimulation
Number analyzed (Participants) | 66
Participants
  No disability | 21
  Mild disability | 26
  Moderate disability | 11
  Marked disability | 6
  Severe disability | 2

47. Secondary Outcome: Global Assessment by Caregiver
Description: as for outcome 44
Time Frame: Day 365
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Stimulation
Number analyzed (Participants) | 70
Participants
  No disability | 25
  Mild disability | 28
  Moderate disability | 11
  Marked disability | 4
  Severe disability | 2

48. Secondary Outcome: Global Assessment by Patient
Description: Global outcome measures are a self-rated questionnaire in which patients assess their own global outcome at each visit
Time Frame: Baseline
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Stimulation
Number analyzed (Participants) | 123
Participants
  No disability | 2
  Mild disability | 3
  Moderate disability | 27
  Marked disability | 59
  Severe disability | 32

49. Secondary Outcome: Global Assessment by Patient
Description: Global outcome measures are a self-rated questionnaire in which patients assess their own global outcome at each visit
Time Frame: Day 90
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Stimulation
Number analyzed (Participants) | 122
Participants
  No disability | 28
  Mild disability | 57
  Moderate disability | 25
  Marked disability | 9
  Severe disability | 3

50. Secondary Outcome: Global Assessment by Patient
Description: Global outcome measures are a self-rated questionnaire in which patients assess their own global outcome at each visit
Time Frame: Day 180
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Stimulation
Number analyzed (Participants) | 118
Participants
  No disability | 35
  Mild disability | 50
  Moderate disability | 21
  Marked disability | 11
  Severe disability | 1

51. Secondary Outcome: Global Assessment by Patient
Description: Global outcome measures are a self-rated questionnaire in which patients assess their own global outcome at each visit
Time Frame: Day 365
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Stimulation
Number analyzed (Participants) | 110
Participants
  No disability | 38
  Mild disability | 45
  Moderate disability | 20
  Marked disability | 6
  Severe disability | 1

52. Secondary Outcome: Subjective Assessment by Patient Since Activation of System
Description: Subjective assessment includes changes in their ET symptoms since the last visit indicated as marked improvement, moderate improvement, mild improvement, worsening, or no change.
Time Frame: Day 90
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Stimulation
Number analyzed (Participants) | 122
Participants
  Marked improvement | 76
  Moderate improvement | 23
  Mild improvement | 8
  Unchanged | 6
  Mild worsening | 7
  Moderate worsening | 0
  Marked worsening | 2

53. Secondary Outcome: Subjective Assessment by Patient Since Activation of System
Description: as for outcome 52
Time Frame: Day 180
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Stimulation
Number analyzed (Participants) | 118
Participants
  Marked improvement | 22
  Moderate improvement | 12
  Mild improvement | 17
  Unchanged | 46
  Mild worsening | 18
  Moderate worsening | 3
  Marked worsening | 0

54. Secondary Outcome: Subjective Assessment by Patient Since Activation of System
Description: as for outcome 52
Time Frame: Day 365
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Stimulation
Number analyzed (Participants) | 109
Participants
  Marked improvement | 17
  Moderate improvement | 13
  Mild improvement | 16
  Unchanged | 45
  Mild worsening | 14
  Moderate worsening | 3
  Marked worsening | 1

55. Secondary Outcome: Number of Participants With Satisfaction With the DBS System's Functioning and Ability to Control Symptoms
Description: At each visit, patients will be asked about their satisfaction with the DBS system's functioning and ability to control symptoms
Time Frame: Day 90
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Stimulation
Number analyzed (Participants) | 122
Participants
  Very Satisfied | 78
  Satisfied | 27
  Indifferent | 7
  Not Satisfied | 3
  Very Unsatisfied | 7

56. Secondary Outcome: Number of Participants With Satisfaction With the DBS System's Functioning and Ability to Control Symptoms
Description: as for outcome 55
Time Frame: Day 180
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Stimulation
Number analyzed (Participants) | 118
Participants
  Very Satisfied | 77
  Satisfied | 28
  Indifferent | 4
  Not Satisfied | 5
  Very Unsatisfied | 4

57. Secondary Outcome: Number of Participants With Satisfaction With the DBS System's Functioning and Ability to Control Symptoms
Description: as for outcome 55
Time Frame: Day 365
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Stimulation
Number analyzed (Participants) | 110
Participants
  Very Satisfied | 76
  Satisfied | 22
  Indifferent | 2
  Not Satisfied | 7
  Very Unsatisfied | 3

58. Secondary Outcome: Number of Participants Who Would Choose to Receive the DBS System Again
Description: At each visit, patients will be asked if they would undergo the DBS procedure again
Time Frame: Day 90
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Stimulation
Number analyzed (Participants) | 122
Participants | 106

59. Secondary Outcome: Number of Participants Who Would Choose to Receive the DBS System Again
Description: At each visit, patients will be asked if they would undergo the DBS procedure again
Time Frame: Day 180
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Stimulation
Number analyzed (Participants) | 118
Participants | 111

60. Secondary Outcome: Number of Participants Who Would Choose to Receive the DBS System Again
Description: At each visit, patients will be asked if they would undergo the DBS procedure again
Time Frame: Day 365
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Stimulation
Number analyzed (Participants) | 110
Participants | 98

61. Secondary Outcome: Number of Participants Who Would Recommend the DBS System
Description: At each visit, patients will be asked if they would recommend the DBS system to others
Time Frame: Day 90
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Stimulation
Number analyzed (Participants) | 122
Participants | 117

62. Secondary Outcome: Number of Participants Who Would Recommend the DBS System
Description: At each visit, patients will be asked if they would recommend the DBS system to others
Time Frame: Day 180
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Stimulation
Number analyzed (Participants) | 117
Participants | 113

63. Secondary Outcome: Number of Participants Who Would Recommend the DBS System
Description: At each visit, patients will be asked if they would recommend the DBS system to others
Time Frame: Day 365
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Stimulation
Number analyzed (Participants) | 100
Participants | 98

64. Secondary Outcome: Beck Depression Inventory II (BDI - II) Score for Depression Symptoms
Description: The Beck Depression Inventory II is A clinical rating scale designed for detecting depression based on the Diagnostic and Statistical Manual of Mental Health Disorders-Fourth Edition (DSM-IV) criteria. This widely used instrument consists of 21 items to assess the intensity of depression in clinical and normal patients. Each item is a list of four statements arranged in increasing severity about a particular symptom of depression. The BDI II questionnaire contains 21 questions, each answer being scored on a scale value of 0 to 3. A score between 0-13 indicates minimal depression, 14-19 mild depression, 20-28 moderate depression and 29-63 severe depression. Total scores are obtained by computing the sum of each score. The scores range from 0 to 63, with higher score indicating greater severity of depressive symptoms.
Time Frame: Baseline
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stimulation
Number analyzed (Participants) | 112
score on a scale | 8.8 (7.6)

65. Secondary Outcome: Change From Baseline in Beck Depression Inventory II (BDI - II) Score for Depression Symptoms
Description: as for outcome 64
Time Frame: Day 365
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stimulation
Number analyzed (Participants) | 112
score on a scale
  Mean Score | 6.8 (7.1)
  Mean Change in Score | -2.0 (6.3)

66. Secondary Outcome: Mini Mental State Exam (MMSE) for Examination of Mental Status
Description: The Mini-Mental State Examination (MMSE) is a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment. It examines functions including registration (repeating named prompts), attention and calculation, recall, language, ability to follow simple commands and orientation. Any score of 24 or more (out of 30) indicates a normal cognition.
Time Frame: Baseline
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stimulation
Number analyzed (Participants) | 110
score on a scale | 29.2 (1.2)

67. Secondary Outcome: Change From Baseline in Mini Mental State Exam (MMSE) For Examination of Mental Status
Description: as for outcome 66
Time Frame: Day 365
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stimulation
Number analyzed (Participants) | 110
score on a scale
  Mean Score | 29.1 (1.4)
  Mean Change in Score | -0.1 (1.2)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Stimulation
All-Cause Mortality (participants affected / at risk) | 3/127
Serious Adverse Events (participants affected / at risk) | 28/127
Other Adverse Events (participants affected / at risk) | 91/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stimulation (N=127)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Cardiac Surgery (Cardiac disorders) | 1 (1)
Myocardiac Infarction (Cardiac disorders) | 1 (1)
Bleeding Gastric Ulcer (Gastrointestinal disorders) | 2 (2)
Death (General disorders) | 3 (3)
Worsening of Pre-Existing Condition (General disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 2 (3)
Septic Shock (Infections and infestations) | 1 (1)
Wound Dehiscence (Injury, poisoning and procedural complications) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Fall With Broken Femur (Musculoskeletal and connective tissue disorders) | 1 (1)
Oesophageal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Intracranial Edema (Nervous system disorders) | 1 (1)
Intracranial Hemorrhage Non Symptomatic (Nervous system disorders) | 1 (1)
Intracranial Hemorrhage Symptomatic Persistant (Nervous system disorders) | 1 (1)
Intracranial Hemorrhage Symptomatic Transient (Nervous system disorders) | 1 (1)
Paresis (Nervous system disorders) | 1 (1)
Right Hemiparesis (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Air Embolism (Surgical and medical procedures) | 1 (1)
Untreated Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stimulation (N=127)
Congestive heart failure (Cardiac disorders) | 1 (2)
Palpitations (Cardiac disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Diabetes (Endocrine disorders) | 1 (1)
Blurred vision left eye (Eye disorders) | 1 (1)
Double vision (Eye disorders) | 2 (2)
Right eye retinal detachment (Eye disorders) | 1 (1)
Visual disturbances (Eye disorders) | 7 (7)
Worsening cataracts (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Decreased taste sensation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Difficulty swallowing (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 5 (5)
Fecal incontinence (Gastrointestinal disorders) | 1 (1)
Gastric reflux (Gastrointestinal disorders) | 1 (1)
Increased dysphagia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Atypical chest pain (General disorders) | 1 (1)
Gait disorder including balance problem (General disorders) | 11 (11)
Head cold (General disorders) | 1 (1)
Heat Intolerance (General disorders) | 1 (1)
Hiccups (General disorders) | 1 (1)
Hoarseness (General disorders) | 2 (2)
Hypophonia (General disorders) | 2 (2)
Jolting or shocking sensations (General disorders) | 17 (18)
Left chest discomfort (General disorders) | 1 (1)
Lightheadedness (General disorders) | 3 (3)
Loss of tremor relief (General disorders) | 1 (1)
Lower extremity edema (General disorders) | 1 (1)
Lower leg cramps at night (General disorders) | 1 (1)
RLE cramping, pain (General disorders) | 1 (1)
Right foot edema (General disorders) | 1 (1)
Right shoulder soreness (General disorders) | 1 (1)
Right thumb triggering (General disorders) | 1 (1)
Sialorrhea (General disorders) | 1 (1)
Sialorrhea - right side of mouth (General disorders) | 1 (1)
Slight worsening of balance (General disorders) | 1 (1)
Tightness, chest (General disorders) | 1 (1)
Tingling in Left arm (General disorders) | 1 (1)
Tooth decay (General disorders) | 1 (1)
Weakness (General disorders) | 2 (2)
Weakness LUE (General disorders) | 1 (1)
Word recall (General disorders) | 1 (1)
Worsening of handwriting (General disorders) | 1 (1)
Flu (Infections and infestations) | 1 (1)
Heavy sinus drainage (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 6 (6)
Left breast abscess (Infections and infestations) | 1 (1)
Left leg edema & cellulitis unrelated to device/surgery (Infections and infestations) | 1 (1)
Left shoulder brusitis (Infections and infestations) | 1 (1)
Burning sensation over implant site (Injury, poisoning and procedural complications) | 1 (1)
DBS system malfunction (Injury, poisoning and procedural complications) | 3 (3)
Dental bridge broke (Injury, poisoning and procedural complications) | 1 (1)
Difficult implant of extensions (Injury, poisoning and procedural complications) | 1 (1)
Drainage from IPG incision line (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Frontal incision erythemic (Injury, poisoning and procedural complications) | 1 (1)
Intermittent stimulation (Injury, poisoning and procedural complications) | 1 (1)
Left Frontal Incision Erythemic (Injury, poisoning and procedural complications) | 1 (1)
Left collor bone fracture from fall (Injury, poisoning and procedural complications) | 1 (1)
Left leg drags when stimulation is on (Injury, poisoning and procedural complications) | 1 (1)
Loss of stimulation (Injury, poisoning and procedural complications) | 6 (6)
Medial Lead Placement Stimulation-Induced Side Effects (Injury, poisoning and procedural complications) | 1 (1)
Mild redness over post-auricular incision (Injury, poisoning and procedural complications) | 1 (1)
Persistent pain at IPG site (Injury, poisoning and procedural complications) | 2 (2)
Post operative discomfort (Injury, poisoning and procedural complications) | 4 (4)
Post operative pain (Injury, poisoning and procedural complications) | 2 (2)
Right arm bruising, hair line fracture (Injury, poisoning and procedural complications) | 1 (1)
Right hip fracture from fall (Injury, poisoning and procedural complications) | 1 (1)
Right hip pain from fall (Injury, poisoning and procedural complications) | 1 (1)
Swelling in area of left extension wire (Injury, poisoning and procedural complications) | 1 (1)
Tenderness around connector site (Injury, poisoning and procedural complications) | 1 (1)
Undesirable changes in stimulation (Injury, poisoning and procedural complications) | 1 (1)
Unsteadiness of right leg when stimulation on (Injury, poisoning and procedural complications) | 1 (1)
Elevated PSA (Investigations) | 1 (1)
Hypercholesterolemia (Investigations) | 1 (1)
Increased heart rate (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diminished appetite (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Bilateral hip pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bilateral leg pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cervical pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dysarthria (Musculoskeletal and connective tissue disorders) | 20 (20)
Dystonia (Musculoskeletal and connective tissue disorders) | 3 (3)
Foot pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Gout (Musculoskeletal and connective tissue disorders) | 2 (2)
Hand/ joint pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Left foot pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Left hip pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Left hip strain (Musculoskeletal and connective tissue disorders) | 1 (1)
Left knee pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Left sciatic leg pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteopenia by bone density scan (Musculoskeletal and connective tissue disorders) | 1 (1)
Right knee pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Tennis elbow (Musculoskeletal and connective tissue disorders) | 1 (1)
Worsening RLS symptoms (Musculoskeletal and connective tissue disorders) | 1 (1)
Worsening of myasthenia gravis (Musculoskeletal and connective tissue disorders) | 1 (1)
Bakers cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Left adnexal cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Aphasia (Nervous system disorders) | 3 (3)
Arm jerks periodically (Nervous system disorders) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Cognitive problems (Nervous system disorders) | 1 (1)
Development of PD symptoms (Nervous system disorders) | 1 (1)
Diminished tremor relief (Nervous system disorders) | 4 (4)
Disequilibrium (Nervous system disorders) | 5 (5)
Dizziness (Nervous system disorders) | 1 (1)
Head tremor (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 12 (13)
Inadequate tremor control (Nervous system disorders) | 1 (1)
Intermittent jerky movement of right hand (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Myoclonic jerks (Nervous system disorders) | 1 (1)
Paresis (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 4 (4)
Postural instability (Nervous system disorders) | 1 (1)
Short term memory problems (Nervous system disorders) | 1 (1)
Spelling difficulty-writes or types words with errors (Nervous system disorders) | 1 (1)
Vivid dreaming (Nervous system disorders) | 1 (1)
Worsened tremor (Nervous system disorders) | 1 (1)
Abnormal thinking (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2)
Confusion (Psychiatric disorders) | 5 (6)
Depression (Psychiatric disorders) | 6 (6)
Hyperinsomnia (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Psychiatric changes (Psychiatric disorders) | 1 (1)
Sleep Walking (Psychiatric disorders) | 1 (1)
Kidney stones (Renal and urinary disorders) | 2 (2)
Urinary Tract infection (Renal and urinary disorders) | 3 (3)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Amenorrhea (Reproductive system and breast disorders) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Intermittent Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Left chest hematoma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Mold allergy resulting in asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema over IPG site (Skin and subcutaneous tissue disorders) | 1 (1)
Multiple skin lesions face, arm, back (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Skin lesion (Skin and subcutaneous tissue disorders) | 3 (3)
Subcutaneous hematoma (Skin and subcutaneous tissue disorders) | 1 (1)
Elective left carpal tunnel release surgery (Surgical and medical procedures) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No